CLINICAL TRIAL: NCT00396175
Title: A Double-Blind, Placebo-Controlled, Multicenter Study To Examine the Effects of Finasteride 1 MG on Serum Prostate-Specific Antigen in Men With Androgenetic Alopecia
Brief Title: Effects of Finasteride on Serum Prostate-Specific Antigen (0906-111)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0906-111; 2006_556
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Finasteride; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0906, finasteride / Duration of Treatment : 48 Weeks
Drug: Comparator : placebo (unspecified) / Duration of Treatment : 48 Weeks

SUMMARY:
A clinical study to collect additional data in order to characterize the reduction in PSA with finasteride 1 mg, and its reversibility in men with androgenetic alopecia between the ages of 40 to 60 years.

ELIGIBILITY:
Inclusion Criteria :

* Men 40 to 60 years of age, and in good general physical and mental health, with androgenetic alopecia

Exclusion Criteria :

* History of previous bladder surgery, acute urinary retention, urethral strictures, repeated urethral catheterizations, repeated urinary tract infections, or active urinary tract infections
* History of treatment with finasteride (PROSCAR or PROPECIA) or hypersensitivity to any component of finasteride.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 355
Dates: Start 1998-03; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Serum Prostatic Specific Antigen (PSA) after 48 weeks of treatment

SECONDARY OUTCOMES:
Reversibility of effects on Serum Prostatic Specific Antigen (PSA) after 24 weeks off drug

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] D'Amico AV, Roehrborn CG. Effect of 1 mg/day finasteride on concentrations of serum prostate-specific antigen in men with androgenic alopecia: a randomised controlled trial. Lancet Oncol. 2007 Jan;8(1):21-5. doi: 10.1016/S1470-2045(06)70981-0. PMID 17196507